CLINICAL TRIAL: NCT06164782
Title: A Survey on Psychosomatic Health Status of Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonggui Yuan (Other)
Responsible Party: Sponsor-Investigator, Yonggui Yuan, Chief of the psychosomatic department, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: CN_Psychosomatic_20231201
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Psychosomatic; Disorder, Multiple; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Pupulation of China: General Pupulation of China

SUMMARY:
A Survey on Psychosomatic Health Status of Chinese Population

DETAILED DESCRIPTION:
This is a nationwide cross-sectional study to investigate psychosomatic symptoms among genral population in China. This study will also focus on the relationship between psychosomatic symptoms and functions and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above;
* Able to complete the scale independently;
* Subjects read informed consent through online questionnaires and agreed to cooperate with relevant assessments.

Exclusion Criteria:

* Individuals with severe physical disease;
* Individuals with cognitive impairment;
* Individuals who cannot finish the online survay independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population in China
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2023-12-17 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychosomatic health status | Baseline
  symptoms severity measured by the symptoms checklist of this study

CONTACTS AND LOCATIONS:
Overall Officials: Yonggui Yuan, Prof., Study Chair — Zhongda Hospital